CLINICAL TRIAL: NCT07203365
Title: Immunogenicity After a Prime Dose and Revaccination With Adjuvanted RSVPreF3 Vaccine in the Most Elderly and Frail Population - an Open-labeled Phase IIIb-trial
Brief Title: RSV Immunogenicity Study in the Elderly (RISE)
Acronym: RISE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karin Karin Loré (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Karin Karin Loré, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RISE; 2024-520141-23-01 (EU CTIS Number)
Record Dates: First submitted 2025-08-22; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: RSV Immunisation
Keywords: RISE; RSV vaccination; Respiratory syncytial virus; Elderly; Arexvy

STUDY DESIGN:
Intervention Model Description: Parallel assignment to evaluate the induction of neutralizing antibodies against RSV A and RSV B following the first dose of Arexvy in two age groups: older adults aged ≥80 years and adults aged 60-65 years.
Masking Description: Not applicable; both arms receive active treatment with the Arexvy vaccine, administered according to the assigned regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals of the age of 60 to 65 years old. (Active Comparator): Participants will receive a prime vaccination with Arexvy (RSV vaccine), followed by a revaccination after one year. These participants will be enrolled at the Clinical Trial Unit at the Academic Specialist Center, Region Stockholm.
  Interventions: Biological: This study examines immune response differences Arexvy between individuals aged 80+ and adults aged 60-65
- Individuals ≥80 years old. (Experimental): Participants will receive a prime vaccination with Arexvy (RSV vaccine) and revaccination after one year. Participants in the older age group (80 years and above) will be enrolled at long-term care facilities at Familjeläkarnas Särskilda boenden (SÄBO).
  Interventions: Biological: This study examines immune response differences Arexvy between individuals aged 80+ and adults aged 60-65

INTERVENTIONS:
Biological: This study examines immune response differences Arexvy between individuals aged 80+ and adults aged 60-65 — The RSV vaccine (Arexvy) has demonstrated efficacy against LRTD over three RSV seasons in individuals aged 60 and older, with an acceptable safety and reactogenicity profile. However, data on vaccine responses in individuals aged 80 and older, including frail individuals, remains limited. This population is particularly affected by severe RSV infections, highlighting the need for further investigation to address these gaps.

SUMMARY:
Respiratory syncytial virus (RSV) is a common cause of respiratory tract infections leading to hospitalizations in infants and in elderly. Arexvy is an approved vaccine for the prevention of RSV infection, however, data on its efficacy in individuals aged 80 years and older remain limited. This study aims to evaluate potential differences in immune responses to Arexvy vaccination between adults aged ≥80 years and those aged 60-65 years.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is a common cause of respiratory tract infections that frequently lead to hospitalization, particularly in infants and older adults. The virus relies on two surface glycoproteins, F and G, for cell fusion and attachment, respectively. Among these, the F protein is the primary target of neutralizing antibodies and a critical focus in RSV vaccine development.

RSV spreads through contaminated nasal secretions via large droplets, primarily transmitted through close human contact or contaminated surfaces. Notably, RSV infection does not confer lasting immunity, and the disease imposes a significant burden on healthcare systems, especially among infants and older adults-particularly those over 75 or with underlying health conditions.

Despite more than half a century of research and a considerable global need, progress in RSV vaccine development has been slow. A key challenge has been inducing antibody (Ab) responses that are sufficiently specific, broad, and long-lasting to provide effective protection. However, in recent years, major strides have been made: two RSV vaccines were approved in 2023, and one in 2024, in both Europe and the United States, for the prevention of lower respiratory tract disease (LRTD) in individuals aged 60 years and older, as well as adults 50-59 years old at increased risk for RSV.

Arexvy, developed and manufactured by GSK, is an adjuvanted RSV vaccine based on the prefusion-stabilized F protein. Its formulation includes the AS01E adjuvant, selected based on prior clinical data. A single dose of Arexvy has demonstrated efficacy against LRTD across three RSV seasons in adults aged 60 and above. The vaccine has shown an acceptable safety and reactogenicity profile.

Despite these advancements, there remains limited data on vaccine responses in individuals aged 80 and above, as well as in frail populations, due to their underrepresentation in ongoing clinical trials. While some immunogenicity data are available, a substantial knowledge gap persists regarding the immune responses elicited by Arexvy in this highly vulnerable group who are disproportionately affected by severe RSV infections. Therefore, studying possible differences in the immune response induced upon vaccination with Arexvy between elderly above 80 years of age and younger individuals (60 65 years old) will provide key insights for defining future vaccination strategies in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals who were born between 1965 and 1960 or 1945 and before, at the time of the first vaccination, who live in the community or in a long-term care facility.
* Individuals who can understand and read Swedish.
* Individuals who can provide written consent and agree (by written consent) to receive the Arexvy vaccine.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Participants who are medically stable in the opinion of the investigator at the time of first vaccination.
* Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate if considered by the investigator as medically stable.

Exclusion Criteria:

* Individuals who are medically immunocompromised, less than 2 years since hematopoietic stem cell transplantation (HSCT) or graft-versus-host disease (GVHD), solid-organ transplanted, using immunosuppressive drugs for treatment of cancer and who have inflammatory mediated or autoimmune conditions, as judged by the Investigator.
* Individuals who have already received an RSV vaccine dose at any time in the past.
* Any known or suspected reaction, hypersensitivity or allergies to be exacerbated by any product or component included in the vaccine and trial.
* Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of participation in the trial.
* Treatment or disease which, according to the investigator, can affect treatment or trial results.
* Any of the following medical conditions: Unstable chronic illness, Recurrent or un-controlled neurological disorders or seizures, Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study, Any other medical condition that in the judgment of the investigator would make intramuscular injection unsafe, Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study, Any history of dementia or any medical condition that moderately or severely impairs cognition and understanding of the informed consent form and/or study procedures, History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Participation in another clinical trial during the study period, or any previous clinical trials with RSV- or hMPV-vaccine or other prophylaxis.
* Planned move during the study period that will prohibit participating in the study until study end.
* Participation of any study personnel or their immediate dependents, family or household members as well as any family relations to Sponsor or PI.
* Co-administration of other vaccines less than 14 days before or after study vaccination. A period of less than 30 days before or after study vaccination applies in the case of Shingrix.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint: | Day 31
  To assess the neutralizing antibody geometric mean titers (GMTs) against RSV A and B one month after the prime dose (day 31) of Arexvy in study participants aged 60-65 years and ≥80 years old, measured by a neutralization assay. Mean geometric increase (MGI), geometric increase (MGI) between day 0 and day 31 after prime will be calculated (equal to the geometric mean of the individual ratio). A more detailed description can be found in section 10.2.1.
Primary objective | Day 31
  To describe the induction of neutralizing antibodies against RSV A and B following the first dose of Arexvy in older adults aged 80 years and older and those aged 60 to 65 years.

SECONDARY OUTCOMES:
Secondary objective: | Between day 0 to 18 month
  To evaluate the reactogenicity of Arexvy by recording the occurrence of solicited adverse events (AEs) in the study participants.
Secondary objectives | Between day 0 to 18 month
  To evaluate the safety of Arexvy in terms of the incidence of unsolicited AEs, SAEs/pIMDs and fatal SAEs.
Secondary endpoint | Between day 0 - 18 month
  Incidence of SAEs, pIMDs, and fatal SAEs among study participants receiving Arexvy.
Seconda y endpoint | Between day 0-day 30 after each vaccination
  Incidence of unsolicited AEs in the study participants with an onset during the 30 day follow-up period after each vaccination.
Secondary endpoint | Between day 0-6 month after each vaccination
  Incidence of SAEs or pIMDs in the study participants from the day of vaccination until 6 months.
Secondary endpoint | Between day 0 to 18 month
  Occurrence of any fatal SAEs from day 1 up to study end.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Hervius Askling, Dr, Principal Investigator — Studieenheten Akademiskt Specialistcentrum; Christian Molnár, Dr, Principal Investigator — Familjeläkarnas Särskilda boenden
Locations (2):
- Sweden (2):
  - Familjeläkarna SÄBO, Saltsjöbaden
  - Akademiskt specialistcentrum Studieenheten, Stockholm

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. However, aggregate study results will be published and reported in accordance with applicable regulations.

DOCUMENTS (2):
  • Study Protocol (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT07203365/Prot_000.pdf
  • Informed Consent Form (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT07203365/ICF_001.pdf